CLINICAL TRIAL: NCT05980195
Title: Cognitive Improvement After cARotid stEnting in HyperBaric Oxygen Therapy Trial (CARE-HBOT)
Brief Title: Cognitive Improvement After Carotid Stenting in Hyperbaric Oxygen Therapy Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CH2023-06-13
Record Dates: First submitted 2023-07-06; First posted 2023-08-07 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Carotid Stenosis; Cognitive Impairment; Hyperbaric Oxygen Therapy; Stent Implantation
MeSH Terms: conditions — Carotid Stenosis; Cognitive Dysfunction | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric oxygen therapy plus standard medical treatment (Experimental): Patients will receive hyperbaric oxygen therapy plus standard medical treatment after stenting
  Interventions: Procedure: Hyperbaric oxygen therapy; Drug: Standard medical treatment; Behavioral: Risk factor management
- Standard medical treatment (Active Comparator): Patients will receive standard medical treatment after stenting
  Interventions: Drug: Standard medical treatment; Behavioral: Risk factor management

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — Hyperbaric oxygen therapy for 30 times within 50 days
  Arms: Hyperbaric oxygen therapy plus standard medical treatment
Drug: Standard medical treatment — Standard medical treatment consists of dual antiplatelet treatment (aspirin 100 mg per day for the entire follow-up, clopidogrel 75 per day mg, or ticagrelor 90 mg twice per day for 3 months after stenting).
  Other Name: Dual antiplatelet therapy for 3 months
Behavioral: Risk factor management — Management of risk factors including hypertension, diabetes, lipoprotein metabolism disorder, smoking and exercise

SUMMARY:
The purpose of CARE-HBOT study is to evaluate whether patients with symptomatic severe carotid artery stenosis with cognitive impairment who underwent hyperbaric oxygen therapy plus standard medical treatment after stent implantation could improve their cognitive function compared with those who underwent standard postoperative medical treatment.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, 1:1 randomized trial. In patients with symptomatic severe carotid artery stenosis with cognitive impairment underwent stent implantation, whether hyperbaric oxygen therapy plus standard medical treatment after stenting could improve their cognitive function compared with those who underwent standard postoperative medical treatment will be studied.

Primary endpoint: Cognitive level at 6 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years
2. National Institute of Health stroke scale (NIHSS) ≤3
3. Culprit vessel was the common carotid artery or extracranial internal carotid artery, involving or not involving the external carotid artery
4. The degree of culprit arterial stenosis is 70-99 % ; based on Digital subtraction angiography (DSA) (According to North American Symptomatic Carotid Endarterectomy Trial (NASCET) method)
5. The diameter of the target vessel between 4.0 mm - 9.0 mm
6. Mini-mental State Examination (MMSE) score : education level-middle school ≤ 24; education level-high school ≤ 20 ; education level-college ≤ 17
7. Baseline modified Rankin Scale (mRS) score ≤ 3
8. Patient understands the purpose and requirements of the study, and has provided informed consent

Exclusion Criteria:

1. Tandem extracranial or intracranial stenosis (70%-99%) or occlusion that is proximal or distal to the target intracranial lesion
2. Serious perioperative complications affecting subsequent hyperbaric oxygen therapy (such as cerebral hemorrhage, disabling stroke, etc.)
3. Any history of brain parenchymal or subarachnoid, subdural or extradural haemorrhage in the past 12 months
4. Hemorrhagic transformation after ischemic stroke within 60 days before enrollment
5. Intracranial artery stenosis caused by non-atherosclerotic lesions, including: arterial dissection, Moyamoya disease, vasculitis disease, herpes zoster, varicella-zoster or other viral vascular diseases, neurosyphilis, any other intracranial infections, any intracranial stenosis related to cerebrospinal fluid cells, radiation-induced vascular disease, fibromuscular dysplasia, sickle cell disease, neurofibromatosis, central nervous system benign vascular disease, postpartum vascular disease, suspected vasospasm, suspicious embolism recanalization, etc
6. Nervous system diseases in the past two years, characterized by transient or fixed neurological deficits (such as partial or secondary generalized seizures of epilepsy, complex or classic migraine, tumor or other intracranial space-occupying lesions, subdural hematoma, brain contusion or other post-traumatic lesions, intracranial infection, demyelinating diseases, intracranial hemorrhage, etc.), which cannot be distinguished from cerebral infarction
7. History of stenting of an intracranial or extracranial artery
8. Presence of any unequivocal cardiac source of embolism
9. Chronic atrial fibrillation; paroxysmal atrial fibrillation or paroxysmal atrial fibrillation in the past 6 months, or a history of paroxysmal atrial fibrillation, requiring long-term anticoagulation
10. Myocardial infarction in the past 30 days
11. Combined with intracranial tumor, aneurysm or intracranial arteriovenous malformation
12. Cannot tolerate dual antiplatelet therapy due to known diseases (such as gastrointestinal bleeding)
13. Contraindications to heparin, aspirin, clopidogrel, ticagrelor, anesthesia, or contrast agents
14. Hemoglobin<100g/L, platelet count <100×109/L, international normalized ratio (INR)>1.5, or heparin-related thrombocytopenia or uncorrectable factors leading to bleeding
15. Not suitable for vessel angiography or endovascular interventional therapy (such as morbid obesity; serious vascular tortuosity that hinders the safe introduction of the guiding catheter)
16. Severe hepatic and renal dysfunction
17. Major surgery within the past 30 days or planned within 90 days
18. Renal artery, iliac artery, and coronary artery requiring simultaneous intervention
19. Life expectancy <1 year
20. Pregnant or lactating women
21. Cognitive assessment and follow-up could not be completed due to factors such as severe aphasia, neuropsychological illness or mental illness or dysarthria and inability to communicate
22. History of drug or alcohol abuse, head trauma or central nervous system infection; current use of drugs that affect cognition
23. Combined with diseases that are not suitable for hyperbaric oxygen therapy (such as untreated pneumothorax, uncontrolled epilepsy, claustrophobia, angle-closure glaucoma, cavitary pulmonary tuberculosis, etc.)
24. Enrollment in another study that would conflict with the current study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 6 months
  Chinese version of Montreal Cognitive Assessment (MoCA) will be use to assess the cognitive level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 30. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | 6 months
  Chinese version of MMSE will be use to assess the cognitive level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 30. Higher scores mean a better outcome.
Auditory Verbal Learning Test (AVLT) | 6 months
  Chinese version of AVLT will be use to assess the cognitive function domain level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 12. Higher scores mean a better outcome.
Symbol Digital Modalities Test (SDMT) | 6 months
  Chinese version of SDMT will be use to assess the cognitive function domain level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 90. Higher scores mean a better outcome.
Digit Span Test (DST) | 6 months
  Chinese version of DST will be use to assess the cognitive function domain level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 22. Higher scores mean a better outcome.
Stroop Color-Word Test (Stroop) | 6 months
  Chinese version of Stroop will be use to assess the cognitive function domain level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 50. Higher scores mean a better outcome.
Trail Making Test (TMT) | 6 months
  Chinese version of TMT will be use to assess the cognitive function domain level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. Recording time consumption. Shorter time consumptions mean a better outcome.
Boston Naming Test (BNT) | 6 months
  Chinese version of BNT will be use to assess the cognitive function domain level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 30. Higher scores mean a better outcome.
Verbal Fluence Test (VFT) | 6 months
  Chinese version of VFT will be use to assess the cognitive function domain level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. Record the number of correct phrases. Higher scores mean a better outcome.
Hamilton Anxiety Scale (HAMA) | 6 months
  Chinese version of HAMA will be use to assess the anxiety level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 64. Higher scores mean a better outcome.
Hamilton Depression Scale (HAMD) | 6 months
  Chinese version of HAMD will be use to assess the depression level of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 96. Higher scores mean a better outcome.
Pittsburgh Sleep Quality Index (PSQI) | 6 months
  Chinese version of PSQI will be use to assess the sleep quality of the hyperbaric oxygen therapy group (HBOT group) and the control group at 6 months after procedure. The minimum value is 0 and the maximum value is 27. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Ma, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolff T, Guirguis-Blake J, Miller T, Gillespie M, Harris R. Screening for carotid artery stenosis: an update of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2007 Dec 18;147(12):860-70. doi: 10.7326/0003-4819-147-12-200712180-00006. PMID 18087057
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Sardar P, Chatterjee S, Aronow HD, Kundu A, Ramchand P, Mukherjee D, Nairooz R, Gray WA, White CJ, Jaff MR, Rosenfield K, Giri J. Carotid Artery Stenting Versus Endarterectomy for Stroke Prevention: A Meta-Analysis of Clinical Trials. J Am Coll Cardiol. 2017 May 9;69(18):2266-2275. doi: 10.1016/j.jacc.2017.02.053. PMID 28473130
- [Background] Kleindorfer DO, Towfighi A, Chaturvedi S, Cockroft KM, Gutierrez J, Lombardi-Hill D, Kamel H, Kernan WN, Kittner SJ, Leira EC, Lennon O, Meschia JF, Nguyen TN, Pollak PM, Santangeli P, Sharrief AZ, Smith SC Jr, Turan TN, Williams LS. 2021 Guideline for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021 Jul;52(7):e364-e467. doi: 10.1161/STR.0000000000000375. Epub 2021 May 24. No abstract available. PMID 34024117
- [Background] Bonati LH, Kakkos S, Berkefeld J, de Borst GJ, Bulbulia R, Halliday A, van Herzeele I, Koncar I, McCabe DJ, Lal A, Ricco JB, Ringleb P, Taylor-Rowan M, Eckstein HH. European Stroke Organisation guideline on endarterectomy and stenting for carotid artery stenosis. Eur Stroke J. 2021 Jun;6(2):I-XLVII. doi: 10.1177/23969873211012121. Epub 2021 May 11. PMID 34414302
- [Background] Sztriha LK, Nemeth D, Sefcsik T, Vecsei L. Carotid stenosis and the cognitive function. J Neurol Sci. 2009 Aug 15;283(1-2):36-40. doi: 10.1016/j.jns.2009.02.307. Epub 2009 Mar 9. PMID 19269651
- [Background] Altinbas A, van Zandvoort MJ, van den Berg E, Jongen LM, Algra A, Moll FL, Nederkoorn PJ, Mali WP, Bonati LH, Brown MM, Kappelle LJ, van der Worp HB. Cognition after carotid endarterectomy or stenting: a randomized comparison. Neurology. 2011 Sep 13;77(11):1084-90. doi: 10.1212/WNL.0b013e31822e55b9. Epub 2011 Aug 31. PMID 21880992
- [Background] Huang P, He XY, Xu M. Effects of Carotid Artery Stent and Carotid Endarterectomy on Cognitive Function in Patients with Carotid Stenosis. Biomed Res Int. 2020 Dec 16;2020:6634537. doi: 10.1155/2020/6634537. eCollection 2020. PMID 33381568
- [Background] Gottfried I, Schottlender N, Ashery U. Hyperbaric Oxygen Treatment-From Mechanisms to Cognitive Improvement. Biomolecules. 2021 Oct 15;11(10):1520. doi: 10.3390/biom11101520. PMID 34680155
- [Background] Hadanny A, Rittblat M, Bitterman M, May-Raz I, Suzin G, Boussi-Gross R, Zemel Y, Bechor Y, Catalogna M, Efrati S. Hyperbaric oxygen therapy improves neurocognitive functions of post-stroke patients - a retrospective analysis. Restor Neurol Neurosci. 2020;38(1):93-107. doi: 10.3233/RNN-190959. PMID 31985478